CLINICAL TRIAL: NCT04178694
Title: The Influence of Non-invasive Ventilation on Metabolism in Healthy Volunteers
Acronym: Ganesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B.U.N. 143201940980
Record Dates: First submitted 2019-11-07; First posted 2019-11-26 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-04

CONDITIONS: Energy Expenditure; Non-invasive Ventilation; Metabolism
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- non-invasive ventilation (Experimental): All subjects will be submitted to non-invasive ventilation with different settings. During the whole period indirect calorimetry will be performed and haemodynamic parameters will be monitored using a non-invasive device. Reversed combined RPE scale will be asked on a regular base.
  Interventions: Device: non-invasive ventilation

INTERVENTIONS:
Device: non-invasive ventilation — non-invasive ventilation will be performed on every subjects

SUMMARY:
Before inclusion in the trial. Careful medical history and medication use will be asked. Once included, 5 healthy subjects non-invasive ventilation(V60, Philips, Eindhoven, The Netherlands) will be administered at a level of positive end expiratory pressure (PEEP) of 4 cmH2O and without additional inspiratory support. Inspiratory support will then increase by 2 cmH2O every 2 minutes until 8 cmH2O is achieved for 2 minutes. The energy expenditure is measured using indirect calorimetry (Q-NRG®, Cosmed, Italy). To measure respiratory effort, the reversed RPE-scale was created for the purpose of the study. It uses the validated "rate of perceived exertion" scale (RPE-scale) which was altered by adding a reversed part. This could result in a score of -10 (no respiratory effort) until +10 ( maximal respiratory effort) where 0 represents the basal respiratory condition. Monitoring of heart rate, blood pressure and cardiac output will be done ( Nexfin®, BMEYE, Amsterdam, The Netherlands).

After termination of the study clinical observation by principal investigator or co-investigator will be done for 15 minutes or until all side effects have worn off. If no side effects are observed, subjects will be released.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* pregnancy
* prisoners
* participation in interventional study in last 2 weeks before enrolment
* Current ongoing disease:
* Cardiac
* respiratory
* ear
* nose
* gastro-intestinal
* neurological
* psychiatric

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | during non-invasive ventilation
  in kcal/day Energy expenditure will be measured using indirect calorimetry during different settings of non invasive ventilation

SECONDARY OUTCOMES:
reversed combined rate of perceived exertion scale | during non-invasive ventilation
  no unit, range: [-10 , +10] based on an existing scale of perceived exertion, a reverse part was added to be able to measure an improvement of respiratory exercise compared to normal state.
respiratory rate | during non-invasive ventilation
  in breaths/min
systolic and diastolic bloodpressure | during non-invasive ventilation
  in mmHg
cardiac output | during non-invasive ventilation
  in liter/min
CO2 production of the body ( VCO2) | during non-invasive ventilation
  in ml/min
O2 consumption of the body (VO2) | during non-invasive ventilation
  in ml/min
Respiratory quotient | during non-invasive ventilation
  no unit

CONTACTS AND LOCATIONS:
Overall Officials: Joop Jonckheer, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No